CLINICAL TRIAL: NCT01916655
Title: Improving the Frequency and Quality of Sleep Apnea Care Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 12-069
Record Dates: First submitted 2013-07-19; First posted 2013-08-05 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Adherence; Chronic Disease; Telemedicine; Continuous Positive Airway Pressure; Mobile Health
MeSH Terms: conditions — Sleep Apnea, Obstructive; Chronic Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (Placebo Comparator): standard and typical PAP (Positive Airway Pressure) educational and support protocol
  Interventions: Behavioral: Usual Care
- Self-Management Care (Experimental): Individualized self-management educational and support protocol
  Interventions: Behavioral: Self-Management Care; Behavioral: Usual Care
- Self-Management Mobile Care (Experimental): Individualized self-management educational and support protocol delivered in part by mobile health tool
  Interventions: Behavioral: Self-Management Mobile Care; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Self-Management Care — Provision of sleep apnea-specific self-management education and support for those who are prescribed CPAP therapy
  Arms: Self-Management Care
Behavioral: Self-Management Mobile Care — Provision of sleep apnea-specific self-management education and support for those who are prescribed CPAP therapy via mobile phone
  Arms: Self-Management Mobile Care
Behavioral: Usual Care — standard and typical CPAP educational and support protocol; is the base level education and support that is provided in the other two interventions in this study.

SUMMARY:
OSA is a major chronic condition affecting the quality of life of millions of Americans. Per the Institute of Medicine new treatment adherence strategies are needed to help improve the quality of care, reduce social and economic costs, and help those with chronic conditions (such as OSA) live healthier and more productive lives through better management of their conditions. Using an mHealth tool to help deliver the investigators' Self-Management intervention and improve the frequency and quality of patient-provider communications is a central component of that discovery process.

DETAILED DESCRIPTION:
The objective of this proposal is to evaluate a new mobile health (mHealth) system for patients with Obstructive Sleep Apnea syndrome (OSA) that facilitates patient-centered, collaborative management for patients prescribed the first-line treatment, continuous positive airway pressure (CPAP). CPAP adherence rates are disappointingly low. The mHealth system proposed for use in the study is informed by the group's previous interventional efforts, including that of an interactive website intervention for OSA patients prescribed CPAP. Limitations of that intervention included use of an immobile desktop computer for website access and that it was not based on a previously evaluated protocol. The advantages to the proposed mHealth system are the use of a mobile device to allow for increased patient-provider communications and the incorporation of the Sleep Apnea Self-Management Program protocol. The evaluative aspect of this proposal is designed as a randomized, controlled clinical trial-Usual Care (control; UC); Self-Management Care (intervention 1; SM); Self-Management via mHealth (intervention 2; SM-Mobile). The key feature of the SM-Mobile intervention is the use of a mHealth tool that allows for the provision of the Self-Management Program through the utilization of audio/visual conferencing, self-monitoring, and treatment tracking with the patient remotely (i.e., in the non-clinic environment).

The overarching aim of the present project is to examine the effect of this patient-centered, collaborative care intervention on improving the quality of care, and increasing CPAP adherence to a clinically meaningful level. The central questions that encompass the conceptual and empirical contours of the study: Does the SM-Mobile intervention have an effect on the patient's experience of care, CPAP adherence, and OSA outcomes relative to Usual Care and Self-Management Care? To answer these research questions, and in the process address fundamental intervention efficacy and cost issues in telemedicine, the proposed randomized, controlled trial aims specifically to achieve the following goals:

This project has the following specific aims:

Aim 1: To examine the effect of the Self-Management Care delivered by mHealth (SM-Mobile) intervention compared to Usual Care (SM) and Self-Management Care (SM) on level of CPAP adherence. The hypothesis is that participants in SM-Mobile group will exhibit higher levels of CPAP adherence compared to the UC and SM groups over the 2-month intervention period.

Aim 2: To examine the effect of the SM-Mobile intervention, compared to Usual Care and Self-Management Care, on the patient's experience of the quality of patient-centered, collaborative care (as measured by the Patient Assessment of Chronic Illness Care and the CAHPS Clinician & Group Survey). The hypothesis is that participants in the SM-Mobile group will experience a greater improvement in patient-centered, collaborative care compared to the UC and SM groups over the 2-month follow-up period.

Aim 3: To examine the effect of SM-Mobile, compared to UC and SM, on OSA apnea outcomes (e.g., OSA symptoms and OSA-specific health-related quality of life [HRQOL]). The hypothesis is that participants in the SM-Mobile group will experience greater improvements in self-reported OSA symptoms and HRQOL from baseline compared to the UC and SM over the 2-month follow-up period.

Aim 4: To perform a basic cost analysis of the SM-Mobile intervention compared to Usual Care, applying a micro-cost methodology of measuring the quantity of inputs used in the production of care and the unit cost of each. This will be a test against the null hypothesis of no significant cost differences between groups.

ELIGIBILITY:
Inclusion Criteria:

The project will have a 4-year timeline. Patients and providers at both the VA Pulmonary Sleep Clinic will participate in this prospective randomized clinical trial. Patients will participate by completing written informed consent, agreeing to be randomized, completing a baseline assessment, participating in the study interventional protocol, and completing follow-up assessments up to one-year post-intervention. The intent is to recruit a study population that is fairly representative of the overall VASDHS population of patients diagnosed with OSA. To this end, inclusion criteria are designed to be as inclusive as possible and are operationalized as follows:

* age > 18 years;
* confirmed diagnosis of OSA;
* being newly prescribed CPAP therapy; and
* having chronic symptoms as noted on screening symptom checklist. OSA diagnosis by the Sleep Clinic has been and is currently consistent with published consensus statements49 that CPAP treatment is indicated when the apnea-hypopnea index (AHI, number of apneas + hypopneas per hour of sleep) is either (1) greater than or equal to 15, or (2) between 5 and 15 AND accompanied by documented sleep apnea symptoms, including excessive daytime sleepiness, impaired cognition, mood disorders, insomnia, and documented cardiovascular diseases. Because mild OSA symptoms are at best modestly correlated with AHI, the research study will focus on patients with moderate to severe sleep apnea, and therefore inclusion criteria will require AHI > 15.

Exclusion Criteria:

* Exclusion criteria include cognitive impairment sufficient to cause inability to complete the protocol (MMSE < 24/30);
* residence in a geographical area outside of San Diego County (which could make some necessary face-to-face contact difficult);
* fatal comorbidity (life expectancy less than 6 months as indicated by treating physician);
* significant documented substance/chemical abuse; or
* other participant circumstances that, in the opinion of a consensus of study team, would interfere with the safety of a prospective participant or their need for treatment (i.e., clinical needs of patient outweighs needs of research study). No exclusion criteria or any other study design elements will be used directly or indirectly to restrict study participation by women, members of minority groups, or primary language. Because men have a greater risk for OSA (and are identified and diagnosed at a greater rate) than women, we anticipate a final sample that reflects the OSA base rate differences on sex. Some minority groups are thought to have higher OSA prevalence rates than Caucasians, so assuming they are being screened/diagnosed at the same rates as Caucasians, we expect minority groups to be included in the study at levels that reflect those rates.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Stepnowsky, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: standard and typical PAP educational and support protocol
  Usual Care: standard and typical CPAP educational and support protocol; is the base level education and support that is provided in the other two interventions in this study.
Period: Overall Study
Arm/Group | Usual Care | Self-Management Care | Self-Management Mobile Care
Started | 131 | 109 | 120
Completed | 116 | 89 | 91
Not Completed | 15 | 20 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Self-Management Care | Self-Management Mobile Care | Total
Number analyzed (Participants) | 131 | 106 | 111 | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (14.0) | 51.7 (13.2) | 54.3 (13.5) | 53.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 13 | 30
  Male | 124 | 96 | 98 | 318
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 6
  Asian | 21 | 16 | 15 | 52
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 3 | 4
  Black or African American | 25 | 20 | 32 | 77
  White | 79 | 68 | 55 | 202
  More than one race | 3 | 0 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 131 | 106 | 111 | 348

OUTCOME MEASURES:

1. Primary Outcome: Positive Airway Pressure Adherence
Description: objective measurement of the amount of time PAP therapy is used at the prescribed pressure
Time Frame: 2 month time point
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Usual Care | Self-Management Care | Self-Management Mobile Care
Number analyzed (Participants) | 131 | 106 | 111
Hours | 3.9 (2.2) | 3.9 (2.4) | 3.8 (2.4)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Usual Care | Self-Management Care | Self-Management Mobile Care
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/89 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/89 | 0/91
Other Adverse Events (participants affected / at risk) | 0/116 | 0/89 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT01916655/Prot_SAP_ICF_000.pdf